CLINICAL TRIAL: NCT03725124
Title: The Lived Experience of Family Planning of Female Patients Diagnosed With Inflammatory Bowel Disease (IBD) and Their Partners During Key Reproductive Stages - a Qualitative Study
Brief Title: Family Planning in Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017GAS97
Record Dates: First submitted 2018-10-29; First posted 2018-10-30 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients: Women with inflammatory bowel disease (IBD.
  Interventions: Other: Interview
- Partners: Partners of women with IBD.
  Interventions: Other: Interview
- Healthcare Professionals: Healthcare professionals working with women with IBD.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Participants will be interviewed on their experience of family planning and inflammatory bowel disease.

SUMMARY:
This study explores the lived experiences of family planning for women with inflammatory bowel disease (IBD) and their partners during the reproductive stages of pre-conception, pregnancy and the postnatal period through qualitative interviews. Insights from existing literature alongside findings from interviews and focus groups with patients and healthcare providers to develop an intervention to address the issues and support needs as identified by study participants.

DETAILED DESCRIPTION:
This study will be conducted in 3 phases:

Phase 1: Literature review (0-9 months). The research literature on pregnancy outcomes and factors affecting family planning decisions of women and men diagnosed with IBD will be systematically searched and reviewed. The findings will be used to prepare a topic guide to be used in the interviews with women and their partners.

Phase 2: Interview study (10-20 months). A topic guide prepared in Phase 1 will provide a structure for in-depth interviews to explore the experience of family planning by women diagnosed with inflammatory bowel disease (IBD) and their partners. Detailed face-to-face interviews will be voice recorded and transcribed verbatim. Each interview may last approximately 45-60 minutes, giving participants sufficient time to share their experience. A total of 24-30 women diagnosed with IBD will be interviewed, where possible selecting 8-10 women at different family planning stages (pre-pregnancy, pregnancy and post-delivery). 3-4 women's partners for in each group, to explore partner's perspective of the pregnancy or pre-conception experience.

Phase 3: Intervention development with focus group interview (21-24 months). The Phase 2 findings will be used to prepare a draft of the intervention to address the issues and support needs as identified by study participants. A group of patients (3-4) and healthcare practitioners (3-4) will be recruited to take part in a joint discussion (focus group interview) on intervention acceptability, and the comments will be used to further develop the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with IBD at different family planning stages (pre-pregnancy, pregnancy and post-partum).
* Women diagnosed with IBD's partners.
* Health practitioners involved with women diagnoses with IBD and on-going care (phase 3 only).

Exclusion Criteria:

* Does not consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women with inflammatory bowel disease (IBD), partners of women with IBD and healthcare professionals working with women with IBD will be recruited via patient groups and secondary care IBD clinics.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Interviews of women with inflammatory bowel disease and their partners to measure their experience and feelings related to fertility and family planning | Up to 14 months
  Exploratory and qualitative in nature with no scale. Experiences of women with inflammatory bowel disease (IBD) and their partners related to fertility and family planning will be sort by interview. Descriptive outcomes will be obtained, but we do not know what they will be until we interview the participants.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, United Kingdom